CLINICAL TRIAL: NCT02427633
Title: A Randomised Controlled Study of the Use of Recovery Positions for Comatose Patients in a Resource Limited Setting
Brief Title: Study of Body Positions in Unconsciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Chittagong Medical College and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BAKMAL1405
Record Dates: First submitted 2015-01-12; First posted 2015-04-28 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Coma
Keywords: recovery position; comatose; resource limited
MeSH Terms: conditions — Coma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Randomized to standard care (control group) - observations only
- UKRC 1997 (Experimental): Randomized to modified UKRC 1997 - Intervention and Observations
  Interventions: Other: Educational Intervention UKRC 1997
- UKRC 2010 (Experimental): Randomized to modified UKRC 2010 - Intervention and Observations
  Interventions: Other: Educational Intervention UKRC 2010

INTERVENTIONS:
Other: Educational Intervention UKRC 1997 — Educational poster intervention indicating the modified UKRC 1997 recovery position
  Arms: UKRC 1997
Other: Educational Intervention UKRC 2010 — Educational poster intervention indicating the modified UKRC 2010 recovery position
  Arms: UKRC 2010

SUMMARY:
In resource limited settings, access to one-on-one nursing care and airway protection by intubation may be unavailable. Patients with coma but adequate oxygenation are frequently cared for on medical wards, and nursed by their family members. The investigators previously audited the use of the recovery position in patients with cerebral malaria and found that its usage was greatly increased by an educational intervention aimed at patient's caregivers. A trend to reduction in coma duration and aspiration pneumonia was also found. Since there is no evidence that placing comatose, non-intubated patients in a recovery position improves outcome, the investigators plan to conduct a randomised controlled study comparing standard care with an educational intervention targeting patients' relatives, teaching them to maintain their relative in one of two different recovery positions. With the preliminary efficacy and safety data and feedback that this study will provide, the investigators would then move to conduct a large multicenter study powered to detect a difference in mortality.

DETAILED DESCRIPTION:
Methods:

In this prospective, three-armed randomised controlled study, patients admitted to the adult medical wards of Chittagong Medical College Hospital with acute onset of reduced consciousness (Glasgow Coma Scale (GCS) <12 for less than 5 days) will be randomised 1:1:1 to one of three arms; standard care (no intervention) or an educational intervention directing placement into one of two recovery positions.

The educational intervention will occur following randomisation and on daily follow-up until recovery from deep coma or death. For patients in the intervention arms, the patients' relatives will be instructed on how to maintain their patient in the recovery position, and an educational poster will be attached to their bed.

Enrolled subjects will be observed 3 times a day until discharge for body position and vital signs including GCS, heart rate, respiratory rate and oxygen saturation.

The primary outcome will be the risk of (hazard ratio) aspiration pneumonia and pneumonitis. The secondary outcome measures will include time to hypoxia, death and coma recovery time. Pulmonary complications will be defined clinically and radiologically. The primary comparison between groups will be the standard care group versus both recovery positions combined. Analysis will be by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Male or female admitted to the medical wards at CMCH
* Current GCS < 12
* Less than 5 day history of reduced consciousness
* Written informed consent obtained through an adult (≥18 years) relative or parent/guardian

Exclusion Criteria:

* Suspected head or spinal injury/trauma requiring appropriate immobilisation and stabilization
* Patient physically restrained by ward staff due to agitation
* Unsuitability for lateral positioning e.g. due to burns on lateral aspects, femoral vascular catheter
* Requirement for nursing in an upright position e.g. due to respiratory insufficiency
* Known or suspected pregnancy
* Intubation
* Patient or family member previously enrolled in this study.
* Consent refused, or no adult (≥18 years) relative or parent/guardian present to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1540 (Actual)
Dates: Start 2014-08-23 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Composite of aspiration pneumonitis or pneumonia | 48 hours after GCS13

SECONDARY OUTCOMES:
Proportion of patients developing hypoxia | 48 hours after GCS13,
Development of pneumonia or pneumonitis, assessed individually | 48 hours after GCS13
Mortality | 7 days post discharge/last follow-up
Time to mortality | 7 days post discharge/last follow-up
Coma recovery time, defined as time to GCS 15 | during hospitalization (defined as time to GCS 15), expected less than 4 weeks
The number of documented episodes of hypoxia | 48 hours after GCS 13
Percentage of observations in the recovery position | whilst GCS<12, expected less than 2 months
Modified Rankin scale | on discharge, expected less than 2 months
Composite of pressure sore, venous thrombosis, arm or leg peripheral nerve or joint injury | whilst GCS<12, expected less than 2 months
Proportion of patients developing a pressure sore | whilst GCS<12, expected less than 2 months
Proportion of patients developing a venous thrombosis, | whilst GCS<12, expected less than 2 months
Proportion of patients developing a new arm or leg peripheral nerve injury | during hospitalization, expected less than 2 months
Proportion of patients developing a new arm or leg joint injury | during hospitalization, expected less than 2 months
Trends in Blood presure | during hospitalization, expected less than 2 months
  measure Systolic and diastolic blood pressure levels
Trends in heart rate | during hospitalization, expected less than 2 months
Proportion of patients developing peripheral venous cannula function | whilst GCS<12, expected less than 2 months
time to hypoxia | 48 hours after GCS13, expected less than 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Kingston, Dr., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Chittagong Medical College Hospital, Chittagong, Bangladesh

REFERENCES:
- [Background] Maude RJ, Hoque G, Hasan MU, Sayeed A, Akter S, Samad R, Alam B, Yunus EB, Rahman R, Rahman W, Chowdhury R, Seal T, Charunwatthana P, Chang CC, White NJ, Faiz MA, Day NP, Dondorp AM, Hossain A. Timing of enteral feeding in cerebral malaria in resource-poor settings: a randomized trial. PLoS One. 2011;6(11):e27273. doi: 10.1371/journal.pone.0027273. Epub 2011 Nov 16. PMID 22110624
- [Background] Koster RW, Baubin MA, Bossaert LL, Caballero A, Cassan P, Castren M, Granja C, Handley AJ, Monsieurs KG, Perkins GD, Raffay V, Sandroni C. European Resuscitation Council Guidelines for Resuscitation 2010 Section 2. Adult basic life support and use of automated external defibrillators. Resuscitation. 2010 Oct;81(10):1277-92. doi: 10.1016/j.resuscitation.2010.08.009. No abstract available. PMID 20956051
- [Background] Resuscitation Council (UK) Resuscitation 2010 Guidelines Edited by Jerry P. Nolan ISBN 978-1-903812-21-1
- [Background] Berg RA, Hemphill R, Abella BS, Aufderheide TP, Cave DM, Hazinski MF, Lerner EB, Rea TD, Sayre MR, Swor RA. Part 5: adult basic life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S685-705. doi: 10.1161/CIRCULATIONAHA.110.970939. PMID 20956221
- [Background] Leopold SJ, personal communication, November 2013.
- [Background] Huxley EJ, Viroslav J, Gray WR, Pierce AK. Pharyngeal aspiration in normal adults and patients with depressed consciousness. Am J Med. 1978 Apr;64(4):564-8. doi: 10.1016/0002-9343(78)90574-0. PMID 645722
- [Background] Adnet F, Baud F. Relation between Glasgow Coma Scale and aspiration pneumonia. Lancet. 1996 Jul 13;348(9020):123-4. doi: 10.1016/s0140-6736(05)64630-2. No abstract available. PMID 8676684
- [Background] Markenson D, Ferguson JD, Chameides L, Cassan P, Chung KL, Epstein JL, Gonzales L, Hazinski MF, Herrington RA, Pellegrino JL, Ratcliff N, Singer AJ; First Aid Chapter Collaborators. Part 13: First aid: 2010 American Heart Association and American Red Cross International Consensus on First Aid Science With Treatment Recommendations. Circulation. 2010 Oct 19;122(16 Suppl 2):S582-605. doi: 10.1161/CIRCULATIONAHA.110.971168. No abstract available. PMID 20956261
- [Background] Adnet F, Borron SW, Finot MA, Minadeo J, Baud FJ. Relation of body position at the time of discovery with suspected aspiration pneumonia in poisoned comatose patients. Crit Care Med. 1999 Apr;27(4):745-8. doi: 10.1097/00003246-199904000-00028. PMID 10321664
- [Background] Turner S, Turner I, Chapman D, Howard P, Champion P, Hatfield J, James A, Marshall S, Barber S. A comparative study of the 1992 and 1997 recovery positions for use in the UK. Resuscitation. 1998 Dec;39(3):153-60. doi: 10.1016/s0300-9572(98)00144-0. PMID 10078804
- [Background] Fulstow R, Smith GB. The new recovery position, a cautionary tale. Resuscitation. 1993 Aug;26(1):89-91. doi: 10.1016/0300-9572(93)90167-o. PMID 8210736
- [Background] Kumar P, Touquet R. Perils of the recovery position: neurapraxia of radial and common peroneal nerve. J Accid Emerg Med. 1996 Jan;13(1):69-70. doi: 10.1136/emj.13.1.69-c. No abstract available. PMID 8821237
- [Background] Rathgeber J, Panzer W, Gunther U, Scholz M, Hoeft A, Bahr J, Kettler D. Influence of different types of recovery positions on perfusion indices of the forearm. Resuscitation. 1996 Jul;32(1):13-7. doi: 10.1016/0300-9572(96)00952-5. PMID 8809913
- [Background] Doxey J. Comparing 1997 Resuscitation Council (UK) recovery position with recovery position of 1992 European Resuscitation Council guidelines: a user's perspective. Resuscitation. 1998 Dec;39(3):161-9. doi: 10.1016/s0300-9572(98)00142-7. PMID 10078805
- [Background] The 1997 Resuscitation Guidelines for use in the United Kingdom April 1997. Resuscitation Council (UK) Publication.
- [Background] Handley AJ, Becker LB, Allen M, van Drenth A, Kramer EB, Montgomery WH. Single rescuer adult basic life support. An advisory statement from the Basic Life Support Working Group of the International Liaison Committee on Resuscitation (ILCOR). Resuscitation. 1997 Apr;34(2):101-8. doi: 10.1016/s0300-9572(97)01099-x. No abstract available. PMID 9141154
- [Background] Handley AJ. Resuscitation. Resuscitation Council (UK) wants everyone who uses new recovery position to report experiences. BMJ. 1997 Nov 15;315(7118):1308. No abstract available. PMID 9390073
- [Background] Guidelines for the Treatment of Malaria. 2nd edition. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK254223/ PMID 25473692
- [Background] Bollig G, Wahl HA, Svendsen MV. Primary school children are able to perform basic life-saving first aid measures. Resuscitation. 2009 Jun;80(6):689-92. doi: 10.1016/j.resuscitation.2009.03.012. Epub 2009 Apr 21. PMID 19386407
- [Background] Stroud M, Duncan H, Nightingale J; British Society of Gastroenterology. Guidelines for enteral feeding in adult hospital patients. Gut. 2003 Dec;52 Suppl 7(Suppl 7):vii1-vii12. doi: 10.1136/gut.52.suppl_7.vii1. No abstract available. PMID 14612488
- [Background] Warner MA, Warner ME, Weber JG. Clinical significance of pulmonary aspiration during the perioperative period. Anesthesiology. 1993 Jan;78(1):56-62. doi: 10.1097/00000542-199301000-00010. PMID 8424572
- [Background] Sakai T, Planinsic RM, Quinlan JJ, Handley LJ, Kim TY, Hilmi IA. The incidence and outcome of perioperative pulmonary aspiration in a university hospital: a 4-year retrospective analysis. Anesth Analg. 2006 Oct;103(4):941-7. doi: 10.1213/01.ane.0000237296.57941.e7. PMID 17000809
- [Background] Lim WS, Baudouin SV, George RC, Hill AT, Jamieson C, Le Jeune I, Macfarlane JT, Read RC, Roberts HJ, Levy ML, Wani M, Woodhead MA; Pneumonia Guidelines Committee of the BTS Standards of Care Committee. BTS guidelines for the management of community acquired pneumonia in adults: update 2009. Thorax. 2009 Oct;64 Suppl 3:iii1-55. doi: 10.1136/thx.2009.121434. No abstract available. PMID 19783532
- [Background] Dalhoff K, Ewig S; Gideline Development Group; Abele-Horn M, Andreas S, Bauer TT, von Baum H, Deja M, Gastmeier P, Gatermann S, Gerlach H, Grabein B, Hoffken G, Kern W, Kramme E, Lange C, Lorenz J, Mayer K, Nachtigall I, Pletz M, Rohde G, Rosseau S, Schaaf B, Schaumann R, Schreiter D, Schutte H, Seifert H, Sitter H, Spies C, Welte T. Adult patients with nosocomial pneumonia: epidemiology, diagnosis, and treatment. Dtsch Arztebl Int. 2013 Sep;110(38):634-40. doi: 10.3238/arztebl.2013.0634. Epub 2013 Sep 20. PMID 24133545
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079